CLINICAL TRIAL: NCT06519955
Title: Peri-incisional Local Infiltration to Improve Pain Control After Periacetabular Osteotomy
Brief Title: Can PLIA Reduce Early Post-operative Pain After PAO Surgery?
Acronym: PILA PAO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael C Willey (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Michael C Willey, Assistant Professor of Orthopedics and Rehabilitation, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202311233
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hip Dysplasia
Keywords: Hip Dysplasia; Periacetabular Osteotomy; PLIA; Peri-Incisional Local Infiltrative Anesthesia
MeSH Terms: conditions — Hip Dislocation | interventions — Ropivacaine; Epinephrine; Ketorolac; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control (No Intervention): No medication administration. Standard of care medications will be offered.
- Post Closure (Active Comparator): Once the fascia has been closed, the PLIA will be administered using a pediatric catheter.
  Interventions: Combination Product: Ropivacaine, Epinephrine, Ketorolac, NaCl (Saline)
- Throughout Procedure (Active Comparator): The injection will be performed throughout the surgical procedure.
  Interventions: Combination Product: Ropivacaine, Epinephrine, Ketorolac, NaCl (Saline)

INTERVENTIONS:
Combination Product: Ropivacaine, Epinephrine, Ketorolac, NaCl (Saline) — Weight 50-74.9 kg:
  * ropivacaine 100mg/epinephrine 50 mcg/ketorolac 15mg in NaCl 0.9% 60mL
  * 2 vials of this for 120mL total
  Weight 75-99.9 kg:
  * Ropivacaine 150mg/epinephrine 100 mcg/ketorolac 15mg in NaCl 0.9% 60mL
  * 2 vials of this for 120mL total
  Weight 100+ kg:
  * Ropivacaine 200mg/epinephrine 150 mcg/ketorolac 15 mg in NaCl 0.9% 60mL
  * 2 vials of this for 120mL total
  Arms: Post Closure; Throughout Procedure

SUMMARY:
The goal of this clinical trial is to compare different peri-incisional local infiltrative anesthesia (PLIA) methods in patients ages 13 to 50 undergoing a periacetabular osteotomy (PAO). The main questions to answer here are:

1. Does PLIA impact post-operative pain after PAO?
2. Does PLIA impact pain medication usage as measured by morphine equivalent dosing (MED) after PAO?
3. Does the timing of PLIA administration impact post-operative pain and MED after PAO? Participants will be asked to complete some surveys; demographics survey, General Self-Efficacy Scale (GSE) and the Pain Resilience Scale. All other information will be gathered from the patients medical chart.

Researchers will compare three groups. 1.) Patients who do not receive PLIA. 2.) Patients who receive PLIA after their incision is closed. 3.) Patients who receive PLIA throughout PAO.

DETAILED DESCRIPTION:
Patients will be approached at their preoperative appointment. This is the only time researchers will conduct study related activities with patients. All other information will be gathered by chart review. Following consent, patients will be asked to complete surveys through REDCap® using a tablet or computer. These include a self-efficacy survey and a grit survey. Patients will then be randomized in a 1:1:1 ratio. 1.) Patients who do not receive PLIA. 2.) Patients who receive PLIA after their incision is closed. 3.) Patients who receive PLIA throughout PAO.

Patients will be blinded to which group they are in, meaning they will not know whether they received the injection or not. Patients may ask to be told what study group they were in at their standard-of-care, 3 month follow-up visit.

Following surgery, patients in all treatment arms will be provided with the same intravenous (patient-controlled analgesia) and oral pain medications scheduled as needed per standard of care.

The research team will review patient medical records to record narcotic use and visual analog scale (VAS) pain scores post-operatively until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or young adult diagnosed with hip dysplasia indicated for PAO at University of Iowa Hospital and Clinics.

Exclusion Criteria:

* Unable to provide informed consent.
* Pregnant or breast-feeding individuals
* Prisoner or ward of the state
* Allergy or medical contradiction to any of the study medications
* Patients undergoing femoral osteotomy or surgical hip dislocation with PAO will be excluded

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain after periacetabular osteotomy. | Post Anesthesia Care Unit (PACU), 24 hours post op
  Severity of pain will be measured by collection of the visual analog scale (VAS) for pain. Scale of 1-10.
Pain medication usage after periacetabular osteotomy. | Post Anesthesia Care Unit (PACU) to end of hospital stay, an average of 3 days.
  The amount of pain medications taken will be measured using morphine equivalent dosing (MED).
The impact of timing of PLIA administration on post-operative pain. | Post Anesthesia Care Unit (PACU) to end of hospital stay, an average of 3 days.
  The mean VAS pain will be compared between the different study groups. Scale of 1-10.
The impact of timing of PLIA administration on MED. | Post Anesthesia Care Unit (PACU) to end of hospital stay, an average of 3 days.
  The mean MED will be compared between the different study groups.

SECONDARY OUTCOMES:
Assessment on depression (PHQ-9) | Preoperative
  A scale to measure depression will be collected to determine the impact on early post-operative pain. Scale of 0-27.
General Self-Efficacy Scale (GSE) | Preoperative
  Scale on self-efficacy will be collected to determine the impact on early post-operative pain. Scale of 10-40
Pain Resilience Scale. | Preoperative
  Scale on pain resilience (grit) will be collected to determine the impact on early post-operative pain. The scale provides two scores, Behavioral Perseverance on a scale of 0-20 and Cognitive/Affective Positivity on a scale of 0-36.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States